CLINICAL TRIAL: NCT04004403
Title: Alternate Day Fasting Combined With Exercise for the Treatment of Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Alternate Day Fasting, Exercise, and NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Krista Varady, Professor of Nutrition, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-0300; R01DK119783 (NIH)
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alternate day fasting (Experimental): These participants will consume 600 kcal on the "fast day" and eat ad libitum at home on alternating "feed days".
  Interventions: Other: Alternate day fasting
- Exercise (Experimental): These participants will participate in a supervised aerobic exercise program 5 times per week, 40-60 min per session, 60-85% HRmax.
  Interventions: Other: Exercise
- Combination alternate day fasting plus exercise (Experimental): These participants will consume 600 kcal on the "fast day" and eat ad libitum at home on alternating "feed days". They will also participate in a supervised aerobic exercise program 5 times per week, 40-60 min per session, 60-85% HRmax.
  Interventions: Other: Alternate day fasting; Other: Exercise
- Control (No Intervention): Controls will be instructed to maintain their weight throughout the trial, and not to change eating or physical activity habits.

INTERVENTIONS:
Other: Alternate day fasting — The diet involves consuming 600 kcal on the "fast day" and eat ad libitum at home on alternating "feed days".
  Arms: Alternate day fasting; Combination alternate day fasting plus exercise
Other: Exercise — The exercise intervention involves supervised aerobic exercise program 5 times per week, 40-60 min per session, 60-85% HRmax.
  Arms: Combination alternate day fasting plus exercise; Exercise

SUMMARY:
Approximately 65% of obese individuals have non-alcoholic fatty liver disease (NAFLD), and this condition is strongly related to the development of insulin resistance and diabetes. Innovative lifestyle strategies to treat NAFLD are critically needed. The proposed research will demonstrate that alternate day fasting (ADF) combined with exercise is an effective non-pharmacological therapy to treat NAFLD.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is characterized by an accumulation of fat in the liver (not resulting from excessive alcohol consumption). Approximately 65% of obese individuals have NAFLD, and this condition is strongly related to the development of insulin resistance and type 2 diabetes. While certain pharmacological agents have been shown to reduce liver fat (i.e. thiazolidinediones), there is mounting concern regarding the safety and weight-gaining effects of these compounds. In light of this, recent research has focused on non-pharmacological lifestyle therapies to reduce hepatic steatosis, such as daily calorie restriction combined with aerobic exercise. Evidence from clinical trials suggest that this combination is an effective lifestyle therapy improve liver fat content and hepatic insulin sensitivity.

More recently, it's been shown that intermittent fasting may produce even greater improvements in hepatic steatosis and hepatic insulin sensitivity, when compared to conventional calorie restriction. For instance, intrahepatic lipid accumulation was lower and insulin sensitivity was higher in mice fasted every other day, when compared to mice who were energy restricted every day. Moreover, data from human trials show that adults with obesity experience greater decreases in insulin and insulin resistance with intermittent fasting versus daily restriction. These findings suggest that intermittent fasting may be a more effective diet therapy to reduce hepatic steatosis and improve insulin sensitivity, when compared to daily calorie restriction. Although these findings are very promising, these data still require confirmation by a randomized controlled clinical trial.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age between 18 to 65 years old
* BMI between 30.0 and 59.9 kg/m2
* NAFLD (hepatic steatosis ≥ 5% confirmed by MRI-PDFF)
* Sedentary (<20 min, 2x/week of light activity at 3-4 metabolic equivalents (METs) for 3 mo prior to study)

EXCLUSION CRITERIA:

* Have chronic liver disease other than NAFLD (hepatitis B or C, primary biliary cirrhosis, sclerosing cholangitis, autoimmune hepatitis, hemochromatosis, Wilson's disease, α1-antitrypsin deficiency)
* Consume excessive amounts of alcohol women: 70 g of ethanol (5 alcoholic drinks per week) and men 140 g of ethanol (10 drinks per week) in the past 6 months)
* Have a history of known cardiovascular, pulmonary or renal disease
* Diagnosed T1DM or T2DM
* Are not weight stable for 3 months prior to the beginning of study (weight gain or loss > 4 kg)
* Are claustrophobic or have implanted metallic/electrical devices (e.g. cardiac pacemaker, neuro-stimulator)
* Are taking drugs that induce steatosis (e.g. corticosteroids, estrogens, methotrexate, Ca channel blockers)
* Are taking drugs that benefit NAFLD (e.g. betaine, pioglitazone, rosiglitazone, metformin, or gemifibrozil)
* Are taking drugs that influence study outcomes (weight loss medications)
* Are perimenopausal or have an irregular menstrual cycle (menses that does not appear every 27-32 days)
* Are pregnant, or trying to become pregnant
* Are smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krista Varady, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alternate Day Fasting | Exercise | Combination Alternate Day Fasting Plus Exercise | Control
Started | 20 | 20 | 20 | 20
Completed | 19 | 15 | 20 | 20
Not Completed | 1 | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adults with obesity and non-alcoholic fatty liver disease
Groups:
- Total: Total of all reporting groups
Arm/Group | Alternate Day Fasting | Exercise | Combination Alternate Day Fasting Plus Exercise | Control | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 20 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (16) | 44 (13) | 44 (13) | 44 (12) | 44 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 17 | 16 | 65
  Male | 4 | 4 | 3 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 1 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 7 | 4 | 24
  White | 10 | 14 | 12 | 13 | 49
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change in Hepatic Steatosis
Description: Hepatic steatosis will be measured by magnetic resonance imaging (MRI-PDFF)
Time Frame: Change from week 1 to week 12
Population: Adults with obesity and NAFLD
Measure: Mean (95% Confidence Interval); unit: liver fat percentage
Arm/Group | Alternate Day Fasting | Exercise | Combination Alternate Day Fasting Plus Exercise | Control
Number analyzed (Participants) | 20 | 20 | 20 | 20
liver fat percentage | -2.25 [-4.46 to -0.04] | -1.3 [-3.8 to 1.2] | -5.48 [-7.77 to -3.18] | -0.17 [-2.17 to 1.83]

2. Secondary Outcome: Change in Body Weight
Description: Measured by digital scale
Time Frame: Change from week 1 to week 12
Population: Adults with obesity and NAFLD
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Alternate Day Fasting | Exercise | Combination Alternate Day Fasting Plus Exercise | Control
Number analyzed (Participants) | 20 | 20 | 20 | 20
kg | -4.45 [-4.93 to -3.97] | -1.79 [-2.33 to -1.26] | -4.18 [-4.65 to -3.71] | -0.52 [-1. to -0.05]

3. Secondary Outcome: Change in Alanine Aminotransferase (ALT)
Description: Measured by a commercial lab (Medstar, Inc)
Time Frame: Change from week 1 to week 12
Population: Adults with obesity and NAFLD
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Alternate Day Fasting | Exercise | Combination Alternate Day Fasting Plus Exercise | Control
Number analyzed (Participants) | 20 | 20 | 20 | 20
U/L | -11.24 [-26.12 to 3.64] | -0.70 [-5.03 to 3.64] | -5.97 [-10.66 to -1.28] | 0.65 [-1.9 to 3.2]

4. Secondary Outcome: Change in Aspartate Aminotransferase (AST)
Description: Measured by a commercial lab (Medstar, Inc)
Time Frame: Change from week 1 to week 12
Population: Adults with obesity and NAFLD
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Alternate Day Fasting | Exercise | Combination Alternate Day Fasting Plus Exercise | Control
Number analyzed (Participants) | 20 | 20 | 20 | 20
U/L | -5.39 [-9.8 to -.98] | .34 [-4.71 to 5.39] | -1.59 [-5.98 to 2.79] | -0.33 [-4.51 to 3.85]

5. Secondary Outcome: Change in Fasting Glucose
Description: Measured by a commercial lab (Medstar, Inc)
Time Frame: Change from week 1 to week 12
Population: Adults with obesity and NAFLD
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Alternate Day Fasting | Exercise | Combination Alternate Day Fasting Plus Exercise | Control
Number analyzed (Participants) | 20 | 20 | 20 | 20
mg/dl | -5.14 [-11.64 to 1.35] | -2.12 [-9.75 to 5.5] | -5.28 [-11.76 to 1.21] | .62 [-5.67 to 6.9]

6. Secondary Outcome: Change in Fasting Insulin
Description: Measured by a commercial lab (Medstar, Inc)
Time Frame: Change from week 1 to week 12
Population: Adults with obesity and NAFLD
Measure: Mean (95% Confidence Interval); unit: uIU/mL
Arm/Group | Alternate Day Fasting | Exercise | Combination Alternate Day Fasting Plus Exercise | Control
Number analyzed (Participants) | 20 | 20 | 20 | 20
uIU/mL | -7.41 [-13.58 to -1.24] | -3.93 [-8.87 to 1.01] | -9.59 [-15.16 to -4.02] | 1.22 [-2.48 to 4.92]

7. Secondary Outcome: Change in Insulin Resistance
Description: Measured by Homeostatic model assessment of insulin resistance (HOMA-IR). The HOMA-IR value was calculated using the formula: [HOMA-IR = glucose (mg/dL) × insulin (mU/L)/405]. Interpretation of HOMA-IR Scores: < 1.0: Normal insulin sensitivity; 1.0-1.9: Mild insulin resistance; > 2.0: Moderate to severe insulin resistance.
Time Frame: Change from week 1 to week 12
Population: Adults with obesity and NAFLD
Measure: Mean (95% Confidence Interval); unit: index
Arm/Group | Alternate Day Fasting | Exercise | Combination Alternate Day Fasting Plus Exercise | Control
Number analyzed (Participants) | 20 | 20 | 20 | 20
index | -1.8 [-3.07 to -.54] | -1.25 [-2.76 to .27] | -2.55 [-4.03 to -1.08] | 0.49 [-0.83 to 1.8]

8. Secondary Outcome: Change in HbA1c
Description: Measured by a commercial lab (Medstar, Inc)
Time Frame: Change from week 1 to week 12
Population: Adults with obesity and NAFLD
Measure: Mean (95% Confidence Interval); unit: percentage of glycosylated hemoglobin
Arm/Group | Alternate Day Fasting | Exercise | Combination Alternate Day Fasting Plus Exercise | Control
Number analyzed (Participants) | 20 | 20 | 20 | 20
percentage of glycosylated hemoglobin | -.12 [-.24 to .01] | .02 [-.13 to .16] | -0.08 [-.2 to .05] | .04 [-0.08 to .16]

ADVERSE EVENTS:
Time Frame: 3 months
Description: The definition of adverse event does not differ from that of of the definitions of clinicaltrials.gov
Arm/Group | Alternate Day Fasting | Exercise | Combination Alternate Day Fasting Plus Exercise | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT04004403/Prot_SAP_000.pdf